CLINICAL TRIAL: NCT06744348
Title: Entire Papilla Preservation Technique in the Treatment of Periodontal Intra-Bony Defects: a One-Year Clinical Follow-Up Study on Its Efficacy and Outcomes
Brief Title: Entire Papilla Preservation Technique in the Treatment of Periodontal IntraBony Defects: a 1-year Follow-up Study
Acronym: EPP
Status: Active, not recruiting | Type: Observational
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Fatma Uçan Yarkaç, assoc. prof, Necmettin Erbakan University
Other Study IDs: 2024/470
Record Dates: First submitted 2024-12-02; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-08

CONDITIONS: Periodontal Diseases; Periodontal Bone Loss
Keywords: microsurgery; clinical attachment level
MeSH Terms: conditions — Periodontal Diseases; Alveolar Bone Loss

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Entire Papila Preservation Tecnique: This innovative approach allows for vertical access to the defect site from the buccal and lingual sides without making incisions in the papillary region. Its goal is to minimize the risk of wound healing failure and the exposure of regenerative biomaterials by fully preserving the interdental papilla over the bony defect
  Interventions: Procedure: ENTİRE PAPİLLA PRESERVATİON

INTERVENTIONS:
Procedure: ENTİRE PAPİLLA PRESERVATİON — The "EPP" technique is a tunnel-like approach of the defect-associated inter-dental papilla. Surgical loupes (3.3× magnification) with LED light illumination were used to increase visibility of the surgical site. Following a buccal intra-crevicular incision, a bevelled vertical releasing incision was performed in the buccal gingiva of the neighbouring inter-dental space and extended just beyond the mucogingival line to provide appropriate mechanical access to the intrabony defect.

SUMMARY:
The aim of this study was to investigate the radiographic and clinical outcomes associated with the whole papilla preservation technique in the treatment of isolated intraosseous defects in patients with stage III periodontitis. The records of 17 systemically healthy patients (12 women and 5 men) diagnosed with stage III periodontitis who underwent the whole papilla preservation technique three months after nonsurgical periodontal treatment were evaluated. The following clinical parameters were recorded at baseline and after treatment: full mouth plaque score (FMPS), full mouth bleeding score (FMBS), probing depths (PD), clinical attachment level (CAL) and gingival recession (GR). The early healing index (EHI) score was assessed 1 week after surgery in both groups. CAL gain was determined as the primary outcome. Baseline data as well as follow-up assessments at 1 month, 3 months, 6 months and 1 year were analyzed to determine the efficacy and long-term outcomes of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* • Systemically healthy individuals.

  * Patients who underwent reconstructive periodontal surgery following the completion of non-surgical treatment.
  * Presence of at least one isolated two- or three-wall intrabony defect with probing depth (PD) ≥7 mm, clinical attachment level (CAL) ≥7 mm and at least 4 mm intrabony component involving predominantly the interproximal area of the affected tooth
  * Full-mouth plaque score (FMPS) and full-mouth bleeding score ≤20%

Exclusion Criteria:

* Individuals who smoke
* Individuals with uncontrolled systemic disease
* Individuals using drugs that affect periodontal tissues
* Individuals during pregnancy and breastfeeding
* Presence of single-walled intraosseous defects
* Flood restoration
* Inadequate endodontic treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The aim of this study was to evaluate the data of 17 systemically healthy patients (12 males and 5 females) aged between 22 and 60 years (mean age 41.5 ± 5.96 years) who underwent a surgical procedure three months after completion of non-surgical periodontal therapy (NSPT).
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2024-07-25 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
PROBİNG DEPTH | 1 YEARS
  Probing Depth (PD) refers to the distance from the gingival margin to the base of the periodontal pocket. It is expressed in mm and a high measurement is a clinically unfavorable value
Clinical Attachment Level | 1 YEARS
  Clinical Attachment Level (CAL) is defined as the distance from the cementoenamel junction (CEJ) to the base of the periodontal pocket. It is expressed in mm and a high measurement is a clinically unfavorable value.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Konya Necmettin Erbakan Üniversitesi, Konya, Meram
  - Konya Necmettin Erbakan Üniversitesi, Konya

IPD SHARING:
Plan to Share IPD: No